CLINICAL TRIAL: NCT03557307
Title: PONENTE: A Multicenter, Open-label, Phase 3b Efficacy and Safety Study of Benralizumab 30 mg Administered Subcutaneously to Reduce Oral Corticosteroid Use in Adult Patients With Severe Eosinophilic Asthma on High Dose Inhaled Corticosteroid Plus Long-acting β2 Agonist and Chronic Oral Corticosteroid Therapy
Brief Title: Study to Evaluate Efficacy and Safety of Benralizumab in Reducing Oral Corticosteroid Use in Adult Patients With Severe Asthma
Acronym: PONENTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3250C00065
Record Dates: First submitted 2018-05-14; First posted 2018-06-15 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Asthma
Keywords: Asthma; Severe Asthma; Oral Corticosteroids
MeSH Terms: conditions — Asthma | interventions — benralizumab

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Benralizumab (Experimental): Benralizumab subcutaneous injection
  Interventions: Biological: Benralizumab

INTERVENTIONS:
Biological: Benralizumab — Benralizumab subcutaneous injection

SUMMARY:
This is a study designed to evaluate efficacy and safety of Benralizumab in reducing the Oral Corticosteroid (OCS) use in adult patients with severe asthma who are receiving OCS with or without additional asthma controller medications.

DETAILED DESCRIPTION:
This is an open-label, multicenter study designed to evaluate efficacy and safety of reducing daily oral corticosteroid (OCS) use after initiation of 30 mg dose of benralizumab administered subcutaneously (SC) in patients with severe eosinophilic asthma receiving high-dose inhaled corticosteroid (ICS)/long-acting β2 agonist (LABA) and OCS with or without additional asthma controller(s).

ELIGIBILITY:
Inclusion Criteria:

1. Peripheral blood eosinophil count of ≥150 cells/μL assessed by central lab at Visit 1 or ≥ 300 cells/μL in the past 12 months
2. History of physician diagnosed asthma requiring continuous treatment with high dose ICS (high-dose ICS is budesonide/formoterol HFA ≥640/18 per day or equivalent, fluticasone propionate DPI > 500/day or equivalent, or authorized generics for these products) plus LABA for at least 6 months prior to Visit 1. The ICS and LABA can be contained within a combination product or given by separate inhalers. The ICS can also be given via nebulized solution for inhalation.
3. Chronic oral corticosteroid therapy equivalent to a daily dose of at least 5 mg of prednisone, for at least 3 continuous months directly preceding Visit 1.
4. Patient should be on a stable OCS dose for at least 4 weeks prior to Visit 1.
5. Non-smokers, current smokers or former smokers with a smoking history of < or =20 pack-years at Visit 1

Exclusion Criteria:

1. Clinically important pulmonary disease other than asthma or ever been diagnosed with pulmonary or systemic disease, other than asthma, that are associated with elevated peripheral eosinophil counts
2. Known history of allergy or reaction to the study drug formulation
3. History of anaphylaxis to any biologic therapy
4. A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with, or has failed to respond to, standard of care therapy
5. Asthma exacerbation requiring use of systemic corticosteroids, or an increase in maintenance dose of OCS, or acute upper/lower respiratory infections requiring antibiotics or antiviral medication within 30 days prior to Visit 2 (first benralizumab dose)
6. A history of known immunodeficiency disorder including history of a positive human immunodeficiency virus (HIV) test
7. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥3 times the upper limit of normal (ULN) confirmed at Visit 1.
8. Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent is obtained
9. Coincident primary adrenal failure (Addison's disease) or irreversible secondary hypoadrenalism due to another independent cause (e.g. pituitary tumour or its treatment)
10. Co-existent inflammatory conditions for which chronic OCS doses are part of their maintenance treatment such as Giant Cell Arteritis, Polymyalgia Rheumatica
11. Exclusion from genetic research may be for any of the exclusion criteria specified in the main study or allogeneic bone marrow transplant, Non-leukocyte depleted whole blood transfusion within 120 days of genetic sample collection
12. Current night-shift workers

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2022-03-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (131):
- United States (23):
  - Research Site, Flagstaff, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Aurora, Colorado
  - Research Site, Newark, Delaware
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Albany, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Normal, Illinois
  - Research Site, Georgetown, Kentucky
  - Research Site, Lakeside Park, Kentucky
  - Research Site, Ann Arbor, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, DuBois, Pennsylvania
  - Research Site, North Charleston, South Carolina
- Argentina (11):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Cap. Fed
  - Research Site, Ciudad Autónoma de Bs. As.
  - Research Site, Ciudad Autónoma de Buenos Aire
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Monte Grande
  - Research Site, Ranelagh
  - Research Site, Rosario
  - Research Site, San Juan Bautista
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Erpent
  - Research Site, Ghent
- Brazil (8):
  - Research Site, Botucatu
  - Research Site, Londrina
  - Research Site, Maringá
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, Santo André
  - Research Site, Sorocaba
  - Research Site, Uberlândia
- Canada (7):
  - Research Site, Vancouver, British Columbia
  - Research Site, Vancouver, CA
  - Research Site, Ajax, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
- Colombia (7):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Cali
  - Research Site, Cartagena
  - Research Site, Floridablanca
  - Research Site, Manizales
  - Research Site, Medellín
- Denmark (4):
  - Research Site, Aalborg
  - Research Site, Herlev
  - Research Site, Hvidovre
  - Research Site, Vejle
- France (9):
  - Research Site, Angers
  - Research Site, Besançon
  - Research Site, Colmar
  - Research Site, Marseille
  - Research Site, Nice
  - Research Site, Orléans
  - Research Site, Reims
  - Research Site, Suresnes
  - Research Site, Tours
- Germany (11):
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Darmstadt
  - Research Site, Frankfurt
  - Research Site, Großhansdorf
  - Research Site, Heidelberg
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Magdeburg
  - Research Site, München
- Italy (8):
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Sassari
  - Research Site, Tradate
- Mexico (6):
  - Research Site, Del. Cuauhtemoc
  - Research Site, Durango
  - Research Site, Guadalajara
  - Research Site, Mérida
  - Research Site, Veracruz
  - Research Site, Villahermosa
- Poland (11):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lubin
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Sosnowiec
  - Research Site, Tarnów
  - Research Site, Wieluń
  - Research Site, Wroclaw
- Russia (6):
  - Research Site, Izhevsk
  - Research Site, Kirov
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Ulyanovsk
- Spain (7):
  - Research Site, Cadiz
  - Research Site, Marbella (Málaga)
  - Research Site, Mérida
  - Research Site, Ourense
  - Research Site, Sant Joan Despí (Barcelona)
  - Research Site, Santiago de Compostela-Coruña
  - Research Site, Zaragoza
- Research Site, Lund, Sweden
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Kaohsiung Hsien
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Yunlin
- United Kingdom (4):
  - Research Site, Bradford
  - Research Site, Cambridge
  - Research Site, London
  - Research Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Menzies-Gow A, Gurnell M, Heaney LG, Corren J, Bel EH, Maspero J, Harrison T, Jackson DJ, Price D, Lugogo N, Kreindler J, Burden A, de Giorgio-Miller A, Faison S, Padilla K, Martin UJ, Garcia Gil E; PONENTE Study Group. Adrenal function recovery after durable oral corticosteroid sparing with benralizumab in the PONENTE study. Eur Respir J. 2022 Dec 22;60(6):2103226. doi: 10.1183/13993003.03226-2021. Print 2022 Dec. PMID 35896216
- [Derived] Menzies-Gow A, Gurnell M, Heaney LG, Corren J, Bel EH, Maspero J, Harrison T, Jackson DJ, Price D, Lugogo N, Kreindler J, Burden A, de Giorgio-Miller A, Padilla K, Martin UJ, Garcia Gil E. Oral corticosteroid elimination via a personalised reduction algorithm in adults with severe, eosinophilic asthma treated with benralizumab (PONENTE): a multicentre, open-label, single-arm study. Lancet Respir Med. 2022 Jan;10(1):47-58. doi: 10.1016/S2213-2600(21)00352-0. Epub 2021 Oct 4. PMID 34619104
- [Derived] Menzies-Gow A, Corren J, Bel EH, Maspero J, Heaney LG, Gurnell M, Wessman P, Martin UJ, Siddiqui S, Garcia Gil E. Corticosteroid tapering with benralizumab treatment for eosinophilic asthma: PONENTE Trial. ERJ Open Res. 2019 Sep 25;5(3):00009-2019. doi: 10.1183/23120541.00009-2019. eCollection 2019 Jul. PMID 31579676
- See also: CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250C00065&attachmentIdentifier=ecf72bab-8195-4bbb-8146-15bdb632a43a&fileName=d3250c00065-csp-v4_Redacted.pdf&versionIdentifier=
- See also: Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250C00065&attachmentIdentifier=c9237f6c-c83b-4019-8b75-9ed31b8fd5d0&fileName=d3250c00065-sap-ed-4-Redacted.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250C00065&attachmentIdentifier=bf47c3cc-9aeb-4c0a-9026-61831356ca8c&fileName=d3250c00065-study-synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 705 participants provided informed consent and were assigned a unique enrollment number prior to screening. Of the 705 patients screened, 598 (84.8%) were eligible to receive Benralizumab 30 mg and entered the study. All 598 (100%) patients received the study drug. 195 of the 538 patients who completed the main study treatment enrolled into PONENTE Long Term Follow Up Substudy.
Pre-assignment Details: In PONENTE, at the first visit, ie, the enrollment visit 1, patients were assigned an enrollment number and then evaluated regarding the protocol mandated inclusion and exclusion criteria. After screening and evaluation, only those eligible to receive Benralizumab 30 mg were assigned treatment and entered a 4 week induction phase on a stable dose of oral corticosteroids (OCS). In Substudy, patients were treated according to healthcare provider discretion with no IP provided by sponsor.
Groups:
- Benra 30 mg: For main study (period 1 (OCS reduction period) and period 2 (maintenance period)): Benralizumab 30 mg administered subcutaneously every 4 weeks. For substudy (period 3 (long term follow up substudy), asthma treatment as per healthcare provider discretion, including Benralizumab 30 mg administered subcutaneously every 4-8 weeks or other biologics.
Period: Period 1: To End of OCS Reduction Phase
Arm/Group | Benra 30 mg
Started (Received study drug) | 598
Completed (Could not reduce OCS dose further according to protocol.) | 563
Not Completed | 35
Not completed — Withdrawal by Subject | 10
Not completed — Adverse Event | 7
Not completed — Protocol Violation | 6
Not completed — Lost to Follow-up | 5
Not completed — other | 3
Not completed — Death | 2
Not completed — Failure to meet inclusion/exclusion criteria | 2
Period: Period 2: Maintenance Phase
Arm/Group | Benra 30 mg
Started (Completed OCS reduction phase.) | 563
Completed (Marked 'Completed' to subject's status on the Disposition CRF) | 536
Not Completed | 27
Not completed — Adverse Event | 4
Not completed — Death | 3
Not completed — Lost to Follow-up | 2
Not completed — Pregnancy | 2
Not completed — Protocol Violation | 11
Not completed — Withdrawal by Subject | 2
Not completed — other | 3
Period: Period 3: Long Term Follow up Substudy
Arm/Group | Benra 30 mg
Started (Patients enrolled in long term follow up substudy) | 195
Asthma Treatment as Per Healthcare Provider Discretion (Treated as per healthcare provider's discretion, including Benra 30 mg administered subcutaneously every 4-8 weeks or other biologics. IP or medications were not provided by the sponsor.) | 195
>=50% Any Biologic (>=50% exposure to any biologic treatment for asthma from the end of maintenance phase of the main study to the Long Term Follow Up visit) | 78
>=50% Benra (>=50% exposure to benralizumab from the end of maintenance phase of the main study to the Long Term follow Up visit, and no previous or concurrent exposure to any other biologic during this period) | 69
Completed | 195
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set
Arm/Group | Benra 30 mg
Number analyzed (Participants) | 598
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (13.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 383
  Male | 215
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race of 9 patients in Full Analysis Set is not recorded.
  Participants
    number analyzed (Participants) | 589
    White | 475
    Black or African American | 26
    Asian | 29
    Native Hawaiian or other Pacific Islander | 1
    American Indian or Alaska Native | 46
    Other | 12

OUTCOME MEASURES:

1. Primary Outcome: Patients Who Achieve 100% Reduction in Daily OCS Dose
Description: Patients who achieve 100% reduction in daily OCS dose that are sustained over at least 4 weeks without worsening of asthma
Time Frame: Baseline to end of OCS reduction phase, an average of approximately 200 days (The duration of the OCS reduction phase may vary based on asthma exacerbations, asthma worsening, HPA integrity , or other safety issues altering the OCS titration schedule.)
Population: Full analysis set - All enrolled patients who received at least one dose of benralizumab are included in the FAS, irrespective of their protocol adherence and continued participation in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Benra 30 mg
Number analyzed (Participants) | 598
Participants | 376
Statistical Analysis 1: Comparison: Benra 30 mg; Test type: Other; Clopper-Pearson Exact CI; One sample Confidence Interval; percentage = 62.9, 95% CI 2-sided [58.86 to 66.76] — Percentage of patients who achieved 100% reduction in daily OCS dose that are sustained over at least 4 weeks without worsening of asthma

2. Primary Outcome: Patients Who Achieve 100% Reduction or a Daily OCS Dose of <=5mg
Description: Patients who achieve 100% reduction or a daily OCS dose of <=5mg, if reason for no further OCS reduction is Adrenal Insufficiency, that are sustained over at least 4 weeks without worsening of asthma
Time Frame: as for outcome 1
Population: All enrolled patients who received at least one dose of benralizumab are included in the FAS, irrespective of their protocol adherence and continued participation in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Benra 30 mg
Number analyzed (Participants) | 598
Participants | 490
Statistical Analysis 1: Comparison: Benra 30 mg; Test type: Other; Clopper-Pearson Exact CI; One sample Confidence Interval; percentage = 81.9, 95% CI 2-sided [78.62 to 84.94] — Percentage of patients who achieve 100% reduction or a daily OCS dose of <=5mg, if reason for no further OCS reduction is Adrenal Insufficiency, that are sustained over at least 4 weeks without worsening of asthma

3. Secondary Outcome: Patients Who Achieve a Daily OCS of ≤5mg
Description: Patients who achieve a daily OCS dose of ≤5 mg (regardless of reason for no further OCS reduction), that are sustained over at least 4 weeks without worsening of asthma
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Benra 30 mg
Number analyzed (Participants) | 598
Participants | 547
Statistical Analysis 1: Comparison: Benra 30 mg; Test type: Other; Clopper-Pearson Exact CI; One sample Confidence Interval; percentage = 91.5, 95% CI 2-sided [88.94 to 93.58] — Percentage of patients who achieve a daily OCS dose of ≤5 mg (regardless of reason for no further OCS reduction), that are sustained over at least 4 weeks without worsening of asthma

4. Secondary Outcome: Patients Who Achieve a ≥90%, ≥75%, and ≥50% Reduction in Daily OCS Dose
Description: Patients who achieve a ≥90%, ≥75%, and ≥50% reduction in daily OCS dose that are sustained over at least 4 weeks without worsening of asthma
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Benra 30 mg
Number analyzed (Participants) | 598
Participants
  ≥90% reduction | 383
  ≥75% reduction | 412
  ≥50% reduction | 489
Statistical Analysis 1: Comparison: Benra 30 mg; Test type: Other; Clopper-Pearson Exact CI; One sample Confidence Interval (≥90% reduction); percentage = 64.0, 95% CI 2-sided [60.06 to 67.90] — Percentage of patients who achieve >=90% reduction in daily OCS dose that are sustained over at least 4 weeks without worsening of asthma
Statistical Analysis 2: Comparison: Benra 30 mg; Test type: Other; Clopper-Pearson Exact CI; One sample Confidence Interval (>=75% reduction); percentage = 68.9, 95% CI 2-sided [65.02 to 72.59] — Percentage of patients who achieve >=75% reduction in daily OCS dose that are sustained over at least 4 weeks without worsening of asthma
Statistical Analysis 3: Comparison: Benra 30 mg; Test type: Other; Clopper-Pearson Exact CI; One sample Confidence Interval (>=50% reduction); percentage = 81.8, 95% CI 2-sided [78.44 to 84.79] — Percentage of patients who achieve >=50% reduction in daily OCS dose that are sustained over at least 4 weeks without worsening of asthma

5. Secondary Outcome: Change From Baseline in Average Daily OCS Dose (mg)
Description: Change from baseline in average daily OCS dose (mg) from start of OCS reduction to end of the OCS reduction phase
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | Benra 30 mg
Number analyzed (Participants) | 593
mg | -8.50 [-9.10 to -7.90]
Statistical Analysis 1: Comparison: Benra 30 mg; Test type: Other; Clopper-Pearson Exact CI; One sample Confidence Interval; percentage change from baseline = -76.92, 95% CI 2-sided [-79.90 to -73.94] — Percentage change from baseline in daily OCS dose at the end of OCS reduction phase

6. Other Pre Specified Outcome: Patients Who Achieve 100% Reduction in Daily OCS Dose From Main Study Baseline OCS Dose to the End of the Long Term Follow up Substudy
Description: as for outcome 1
Time Frame: from main study baseline to the end of the long term follow up substudy, an average of approximate 922 days.
Population: Long term follow up analysis set - All patients who enrolled in Long Term Follow Up substudy
Measure: Count of Participants; unit: Participants
Groups:
- Asthma Treatment as Per Healthcare Provider Discretion: Treated as per healthcare provider's discretion, including Benra 30 mg administered every 4 to 8 weeks or other biologics. IP or medications were not provided by the sponsor.
- >=50% Any Biologic: >=50% exposure to any biologic treatment for asthma from the end of maintenance phase of the main study to the Long Term Follow Up visit
- >=50% Benra: >=50% exposure to benralizumab from the end of maintenance phase of the main study to the Long Term follow Up visit, and no previous or concurrent exposure to any other biologic during this period
Arm/Group | Asthma Treatment as Per Healthcare Provider Discretion | >=50% Any Biologic | >=50% Benra
Number analyzed (Participants) | 195 | 78 | 69
Participants | 138 | 60 | 54

7. Other Pre Specified Outcome: Patients Who Achieve a Daily OCS Dose of ≤5 mg at the End of the Long Term Follow up Substudy
Description: as for outcome 3
Time Frame: from main study baseline to the end of the long term follow up substudy, an average of approximate 922 days.
Population: Long Term Follow Up analysis set - All patients who enrolled in Long Term Follow Up substudy
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma Treatment as Per Healthcare Provider Discretion | >=50% Any Biologic | >=50% Benra
Number analyzed (Participants) | 195 | 78 | 69
Participants | 177 | 72 | 65

8. Other Pre Specified Outcome: Patients Who Achieve ≥90%, ≥75%, ≥50% or >0% OCS Reduction From Main Study Baseline OCS Dose to the End of the Long Term Follow up Substudy
Description: as for outcome 4
Time Frame: from main study baseline to the end of the long term follow up substudy, an average of approximate 922 days.
Population: Long Term Follow Up analysis set - All patients who enrolled in Long Term Follow Up substudy
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma Treatment as Per Healthcare Provider Discretion | >=50% Any Biologic | >=50% Benra
Number analyzed (Participants) | 195 | 78 | 69
Participants
  >=90% reduction | 141 | 61 | 55
  >=75% reduction | 151 | 64 | 58
  >=50% reduction | 172 | 71 | 64
  >0% reduction | 175 | 72 | 65

9. Other Pre Specified Outcome: Change in Daily OCS Dose (mg) From Main Study Baseline to the End of the Long Term Follow up Substudy
Description: Change in average daily OCS dose (mg) from main study baseline to the end of the long term follow up substudy
Time Frame: from main study baseline to the end of the long term follow up substudy, an average of approximate 922 days.
Population: Long Term Follow Up analysis set - All patients who enrolled in Long Term Follow Up substudy
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | Asthma Treatment as Per Healthcare Provider Discretion | >=50% Any Biologic | >=50% Benra
Number analyzed (Participants) | 195 | 78 | 69
mg | -10.01 [-11.26 to -8.76] | -10.28 [-12.16 to -8.41] | -10.8 [-12.85 to -8.75]

ADVERSE EVENTS:
Time Frame: Main study: From first dose of study drug until end of study, with an average of 405 days. Substudy: on-study period, between the date of informed consent for the substudy and the last available visit or contact for a patient, with an average of 18 days.
Groups:
- Benra 30 mg: For main study (period 1 (OCS reduction period) and period 2 (maintenance period)): Benralizumab 30 mg administered subcutaneously every 4 weeks.
Arm/Group | Benra 30 mg | Asthma Treatment as Per Healthcare Provider Discretion | >=50% Any Biologic | >=50% Benra
All-Cause Mortality (participants affected / at risk) | 5/598 | 0/195 | 0/78 | 0/69
Serious Adverse Events (participants affected / at risk) | 89/598 | 0/195 | 0/78 | 0/69
Other Adverse Events (participants affected / at risk) | 181/598 | 0/195 | 0/78 | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg (N=598) | Asthma Treatment as Per Healthcare Provider Discretion (N=195) | >=50% Any Biologic (N=78) | >=50% Benra (N=69)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemophilus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 11 (11) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apallic syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast calcifications (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspirin-exacerbated respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 23 (33) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic rhinosinusitis with nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism arterial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg (N=598) | Asthma Treatment as Per Healthcare Provider Discretion (N=195) | >=50% Any Biologic (N=78) | >=50% Benra (N=69)
Influenza like illness (General disorders) | 33 (34) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 64 (92) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 19 (22) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 25 (28) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 28 (31) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 29 (38) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 21 (21) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
During COVID-19 pandemic, for ongoing patients, patient dosing, and scheduled visits are inevitably impacted, but the primary endpoint was not impacted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
≥ 60 days prior to submission of material for publication/presentation, Institution and PI shall jointly provide AZ with material for review. No publication/presentation may include any of AZ's Confidential Information without AZ's written approval. AZ can request Inst. and PI to withhold material from submission for publication/presentation for an additional 90 days to allow AZ to establish and preserve its proprietary rights in the material being submitted for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2020-10-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT03557307/Prot_008.pdf
  • Statistical Analysis Plan (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT03557307/SAP_009.pdf